CLINICAL TRIAL: NCT04763278
Title: Validation of User Needs of the Point Digit With Partial Hand Amputees
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Point Designs (Industry)
Collaborators: University of Colorado, Denver (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 253922; R42HD097827 (NIH)
Record Dates: First submitted 2021-02-15; First posted 2021-02-21 (Actual); Results first posted 2024-09-27 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-09

CONDITIONS: Amputation; Traumatic, Hand

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Prosthesis (Experimental): Patient is temporarily fit with Point Digit partial hand prosthetic system
  Interventions: Device: Point Digit

INTERVENTIONS:
Device: Point Digit — The Point Digit partial hand prosthetic system consists of 1-4 ratcheting mechanical digits and a mounting bracket

SUMMARY:
The objective of the device feasibility study will be to validate the user needs of the Point Digit system. This study will be a single group intervention model where one group of 5 partial hand amputees will be asked to perform several tasks. Successful completion of a task results in a fulfilled user need. Failure to complete a task results in an unfulfilled user need.

ELIGIBILITY:
Inclusion Criteria:

* Partial hand amputees with absence of index and/or middle fingers and presence of thumb. Additional finger loss is acceptable if all other criterion are met.
* Fluent in English
* Individuals aged 18 or greater

Exclusion Criteria:

* Significant cognitive deficits as determined upon clinical evaluation
* Significant neurological deficits as determined upon clinical evaluation
* Significant physical deficits of the residual limb impacting full participation in the study as determined upon clinical evaluation
* Uncontrolled pain or phantom pain impacting full participation in the study as determined upon occupational therapist evaluation
* Serious uncontrolled medical problems as judged by the project therapist.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2021-01-07 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-03-30 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Denver | Anschutz Medical Campus, Aurora, Colorado
  - Point Designs, Lafayette, Colorado

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Prosthesis
Started | 7
Completed | 7
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 3
  More than one race | 0
  Unknown or Not Reported | 4

OUTCOME MEASURES:

1. Primary Outcome: VAL-1: System Comfort Validation Test
Description: User wears Point Digit(s) for a full day (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall be comfortable for a full day's use. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (8 hours)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

2. Primary Outcome: VAL-2: Unilateral Function Validation Test
Description: User flexes and extends the Point Digit(s) without using contralateral hand (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall allow the user to flex and extend finger without their second hand. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

3. Primary Outcome: VAL-3.1: System Robustness Validation Test With 25 lb Bag
Description: User lifts a 25 lb. bag with Point Digit(s) (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall be robust enough to operate in challenging environments. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

4. Primary Outcome: VAL-3.2: Robustness Validation Test With Hammer
Description: User grips a hammer with Point Digit(s) and drives a nail into a piece of wood (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall be robust enough to operate in challenging environments. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

5. Primary Outcome: VAL-4: Object Release Validation Test
Description: User releases Point Digit(s) while performing an active grasp by pressing the dorsal button (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall be releasable while performing active grasps. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

6. Primary Outcome: VAL-5: Position Function Validation Test
Description: User positions Point Digit(s) into each of the locking positions (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall have a smooth ratcheting mechanism. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

7. Primary Outcome: VAL-6: Extension Function Validation Test
Description: User activates spring-back mechanism by using (1) contralateral hand, (2) tabletop, and (3) side or thigh (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall have a reliable auto spring-back mechanism. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

8. Primary Outcome: VAL-7: Grip Functions Validation Test
Description: User grips a 5 lb. cylindrical smooth object using Point Digit(s) for 10 seconds (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall have high grip surface friction. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

9. Primary Outcome: VAL-8: Fine Motor Function Validation Test
Description: User picks up 1 coin from a smooth tabletop (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall have a pronounced fingernail. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (10 minutes)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

10. Primary Outcome: VAL-9: Overall Function & Robustness Validation Test
Description: User performs VAL-1 through VAL-8 (Pass/Fail). This validation method was used to confirm the following user need of the Point Digit has been met: Point Digit shall be robustly attached to mounting system. A simple pass/fail result was recorded for each user need for each participant. An overall passing rate above 80% across all user needs and participants is considered a success. Each participant attended a single-day experimental session. A day-use prosthetic socket was fabricated and Point Digits were mounted to the socket. Then, each participant attempted the validation test.
Time Frame: Day 1 (8 hours)
Measure: Number; unit: % of participants who Passed test
Arm/Group | Prosthesis
Number analyzed (Participants) | 7
% of participants who Passed test | 100

ADVERSE EVENTS:
Time Frame: an average of 1 day
Arm/Group | Prosthesis
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol (2019-03-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT04763278/Prot_000.pdf